## A cluster randomized controlled trial of an after-school playground curriculum intervention to improve children's physical, social, and emotional health: Study protocol for the PLAYground project

NCT ID not yet assigned

Date: June 20, 2022

## **Informed Consent: Child Assent**

| I have been told that my mom or dad has said it's okay for me to take part in a project about movement and activity in my afterschool program. |
|---|
| I will wear a physical activity monitor on my wrist, like a watch, for seven days. I will also complete a survey that will take about five or ten minutes. |
| I am taking part because I want to. I know that I can stop at any time if I want to and it will be okay if I want to stop. |
| I know that I can ask my teachers or the ASU research team about the study at any time if I do not understand something. |
| Your Name Date |

## **Informed Consent: Parent Consent**

Our names are Dr. XXX and Dr. XXX and we are professors at XXX University in the College of XXX and XXX College. We are conducting a research study to learn about social and emotional development through physical activity, and student leadership in recess activities.

We are inviting your child's participation, which will involve wearing a small physical activity monitor on their wrist each day for one week twice a year. The monitor is made by Actigraph and measures your child's level of movement. Your child would put the monitor on when they arrive at the Xplore afterschool program and wear it for one full week. There is no need to charge the device, as the battery lasts for several weeks. Your child can comfortably wear the device at all times, except when swimming. Your child will wear the device two times during the year - once in the fall and once in the spring. After returning the device at the end of each week, your child will receive a \$10 gift card. Your child will also be asked to complete a 5-10-minute survey related to their participation in the Xplore after school program and serving as a recess leader twice a year. In addition, demographic information will be collected (i.e., age, gender, ethnic background). Your child may also be asked to participate in a short (15 minute) interview twice a year.

School level data will be collected including attendance records and behavior referrals; however, this will not include specific information for your child. This information is being collected in order to determine if the changes in the afterschool program lead to school level positive changes in attendance and fewer behavioral referrals.

Your child's participation in this study is voluntary. If you choose not to have your child participate or to withdraw your child from the study at any time, there will be no penalty and it will not affect their grade or experience at school. Likewise, if your child chooses not to participate or to withdraw from the study at any time, there will be no penalty. The results of the research study may be published, but your child's name will not be used.

The direct benefits to your child include learning about how to lead games on the playground to promote inclusion, social and emotional health, and physical activity. Further, all children will receive leadership training to promote playground activities during recess at their school. There are no risks to participating in the project as activities will be integrated into the regular Xplore program. Again, the results of this study may be used in reports, presentations, or publications but your child's name will not be known or used.

If you have any questions concerning the research study or your child's participation in this study, please email us at XXX.

| Sincerely, |
|-----------------------------------------|
| xxx |
| *************************************** |

| By signing below, you are giving correturn to your child's Xplore progran | he above study. Please | |
|---|---|---|
| Child's Name | Child's Teacher | |
| Parent Signature | Parent Printed Nam | ne Date |
| program and during recess to use | I videos of students engaged in the X in newspaper or research articles or ermission to use pictures and videos | presentations. By |
| Parent Signature | Parent Name | Date |

If you have any questions about you or your child's rights as a subject/participant in this research, or if you feel you or your child have been placed at risk, you can contact the Chair of the Human Subjects Institutional Review Board, through the Office of Research Integrity and Assurance, at XXX.

Dear Healthy School Leader:

Our names are Dr. XXX and Dr. XXX and we are professors at XXX University in the College of XXX and XXX College. We are conducting a research study to learn about social and emotional development through physical activity, and student leadership in recess activities.

We are inviting your participation as a research participant in our project. This will involve participating in a training to promote social and emotional learning through physical activity. As a healthy school teacher at your school, you will be asked to complete a 5-10-minute survey about your perceptions of changes during recess twice a year. We will also ask you to complete observations of children during recess. The observations will take 5-10 minutes twice a year. You may also be asked to participate in an interview (30 minutes) twice a year. Specifically, we can use your answers to further improve and/or draw conclusions about how to make recess programs more effective in developing both social and emotional learning and physical activity patterns as well as to make these more sustainable in the future. In exchange for your participation, you will receive a \$50 gift card each semester.

Only the researchers will have access to your data. The data will be protected and remain confidential. Your participation in this study is voluntary and you may choose to withdraw at any time. If you choose not to not participate or withdraw from the study there will be no penalty and it will not affect your job status. Data collection will take place during the fall and again in the spring.

The direct benefits to you include gaining knowledge to promote social and emotional learning and physical activity during recess to help children lead healthier lives.

There are no foreseeable risks or discomforts to your participation in training and completing surveys. During survey completion you do not have to answer any question that you do not want to. Your responses will also remain confidential. The results of this study may be used in reports, presentations, or publications but your name will not be known.

If you have any questions concerning the research study or your participation in this study, please call me at.

| Sincerely,<br>XXX | | |
|---|---|---|
| By signing below, you a | re giving consent for your participa | ation in the above study. |
| Signature | Name | Date |
| program and recess to | use in newspaper or research a | students engaged in the after-school rticles or presentations. By signing below, f you in the after-school program and during |
| Signature | <br>Name | <br>Date |

If you have any questions about your rights as a subject/participant in this research, or if you feel you

| have been placed at risk, you can contact the Chair of the Human Subjects Institutional Review Board, through the Office of Research Integrity and Assurance, at XXX. |
|---|